CLINICAL TRIAL: NCT04221763
Title: Evaluation of Mechanisms and Innovations in Cardiac Resynchronization Therapy
Brief Title: Mechanisms and Innovations in Cardiac Resynchronisation Therapy
Acronym: MIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18HH4801; FS/19/4/34013 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2019-11-04; First posted 2020-01-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Left Ventricular Systolic Dysfunction; Left Bundle-Branch Block; Right Bundle-Branch Block; Non-Specific Intraventricular Conduction Defect
Keywords: Cardiac resynchronization therapy; His bundle pacing; Haemodynamics; ECGI
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Bundle-Branch Block | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: 60 patients with heart failure, severe left ventricular systolic dysfunction and cardiac conduction abnormality (QRS > 120ms) will be recruited and undergo an attempt at His bundle, left bundle pacing and biventricular pacing. Patients will have acute haemodynamic and electrical measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Heart failure and abnormal cardiac conduction (Experimental): Subjects will have an attempt at His-bundle pacing, left bundle pacing and biventricular pacing. Pacing at the His bundle and the left bundle will be attempted using a Medtronic SelectSecure™, Model 3830 lead. Delivery of the lead utilizes a deflectable sheath, the Medtronic SelectSite™, Model C304. Biventricular pacing will utilise a left ventricular lead placed in the coronary sinus using any of the 5 manufactures of CS leads Biotronik, Boston Scientific, Medtronic, Sorin, and St. Jude Medical or in participants receiving permanent conduction system pacing left ventricular pacing will be achieved using a Cordis ATW™ wire placed in the coronary sinus.
  Interventions: Device: His-bundle pacing.

INTERVENTIONS:
Device: His-bundle pacing. — Cardiac resynchronisation therapy can be achieved using biventricular pacing involving placement of three leads into the right atrium, right ventricle and coronary sinus (epicardial left ventricle). Alternatively the third lead may be placed at the bundle of His or left ventricular septum to pace the left bundle directly.
  Other Names: Left bundle pacing; Biventricular pacing; Combined His-bundle and left ventricular epicardial pacing (HOT-CRT)

SUMMARY:
The aim of this study is to compare the effectiveness of multiple modalities of cardiac resynchronisation therapy using high precision acute electrical and haemodynamic measurements.These modalities include biventricular pacing and conduction system pacing utilising His bundle and left bundle pacing. Conduction system pacing is a more physiological form of pacing. The study hypothesises that this will produce more effective cardiac resynchronisation.

DETAILED DESCRIPTION:
This is a single centre acute electrical/haemodynamic and observational study of a subgroup of patients with heart failure. A total of 60 will be recruited. The acute study involves within patient comparison of biventricular and conduction system pacing using detailed electrical mapping and high precision haemodynamic measurement protocol.

Participants will have permanent conduction system pacing if;

* Baseline left bundle branch block and QRS > 140ms or QRS >150ms and any QRS morphology AND
* Conduction system pacing is successful at reducing QRS duration by 20ms or more with satisfactory pacing parameters.

Participants who receive permanent conduction system pacing will have follow up at 6 weeks, 3 months, 6 months and 12 months. Non-invasive markers including mechanical activation pattern (echocardiography and cardiac MRI) and electrical activation pattern (ultra-high frequency electrocardiography) will be used to identify the characteristics of patients who benefit from conduction system pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for conventional CRT
* Severe heart failure (LVEF, a measure of heart pumping, < 35% - severe)
* Prolonged QRS duration (>120ms)
* Adults willing to take part (age > 18 years)
* Able to give consent

Exclusion Criteria:

* Unable to give consent
* Children (age < 18 years)
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Acute change is systolic blood pressure | 20 minutes
  Mean change in systolic blood pressure (mmHg) from atrial pacing to AV sequential CRT pacing (HBP, LBP, epiBVP and combined HPB with epiLVP) at optimal AV delay measured in mmHg.
Acute electrical measurements | 20 minutes
  Mean change in left ventricular activation time (Milliseconds) (measured using ECGI) during AV sequential CRT pacing (HBP, LBP, epiBVP and combined HPB with epiLVP) at optimal AV delay measured in Milliseconds.

SECONDARY OUTCOMES:
Conduction system battery longevity | 6 weeks, 3 months, 6 months, 12 months.
  The measurements include battery longevity measured in months.
Conduction system lead threshold | 6 weeks, 3 months, 6 months, 12 months.
  The measurements include lead threshold to achieved QRS narrowing measured in Volts at 0.5ms and 1ms.
Heart failure symptoms | 6 months
  Heart failure symptoms of patients with permanent conduction system leads will be assessed at follow up at 3 month, 6 months and 12 months. The symptoms will be assessed using the Minnesota living with heart failure questionnaire score.
Left ventricular ejection fraction | 12 months
  Patients with permanent conduction system leads will undergo a repeat echocardiography and measure their left ventricular ejection fraction.
Cardiopulmonary exercise testing | 6 months
  Patients with permanent conduction system leads will undergo symptom assessment with a repeat cardio-pulmonary exercise test to measure MVO2 in litres/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Whinnett, BM BS B, Study Chair — Imperial College London
Locations (1):
- Hammersmith Hospital Imperial College NHS trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the electrical data obtained from non-invasive electrical mapping with Medtronic (industry company)
Supporting Information: Analytic Code
Time Frame: 3 years
Access Criteria: Medtronic will only have access to anonymised data in the form of non-invasive electrical maps (ECGi, CardioInsight)

REFERENCES:
- [Background] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Background] Vijayaraman P, Herweg B, Ellenbogen KA, Gajek J. His-Optimized Cardiac Resynchronization Therapy to Maximize Electrical Resynchronization: A Feasibility Study. Circ Arrhythm Electrophysiol. 2019 Feb;12(2):e006934. doi: 10.1161/CIRCEP.118.006934. PMID 30681348